CLINICAL TRIAL: NCT02994017
Title: Prognostic Value of Functional Exercise Test (EFX) in Cystic Fibrosis
Acronym: EFX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011_31; 2011-A01532-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-08-16; First posted 2016-12-15 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; Cardiopulmonary exercise testing; prognostic
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cystic fibrosis patients (Other)
  Interventions: Other: cardiopulmonary exercise testing

INTERVENTIONS:
Other: cardiopulmonary exercise testing — The Cardiopulmonary exercise testing (CPET) was performed at the beginning of the study, the same at each center. Each patient underwent a symptom-limited incremental exercise test on an ergometric bicycle (Ergoline-Ergometrics 800®). The protocol included a warm-up period of 3 min at 20 W followed by a progressively increasing work rate (WR) in a ramp fashion and then 3 min recovery. The ramped WR increment was individualized (range,8-30 W/min). during exercise, heart rate (HR) was monitored continuously by 12-lead ECG, and arterial oxygen saturation (SpO2) was measured by pulse oximetry (Nellcor N-395). The expired gases were analyzed with an Ergocard®, focusing on oxygen consumption(VO2), carbon dioxide production (VCO2), minute ventilation (VE), and tidal volume (VT).

SUMMARY:
The objective of study is to prospectively determine if CPET with blood gas analysis should have a prognostic value in CF. The study plans to include 300 cystic fibrosis patients. Inclusion criteria will be: age >15 years, cystic fibrosis confirmed by chloride sweat test or genetic analysis, clinical and functional stability in the 2 month before CPET. Patients will perform a maximal exercise test on a cycloergometer during the inclusion visit, with pulmonary function testing and a six-minute walk test. The study will also include a visit every 6 months with: body mass index calculation, pulmonary function testing with DLCO (diffusing lung capacity for carbon monoxide), a six minute walk test, and antibacteriological study of sputum. The results of this study could help identify earlier the patients for referral to a lung transplantation centre, by using the usual criteria and the CPET abnormalities.

DETAILED DESCRIPTION:
Current guidelines for referring cystic fibrosis (CF) patients for lung transplantation, based on clinical and functional resting parameters, are insufficient to predict 3-year mortality. Previous studies have shown that sex, impaired pulmonary function, undernutrition and colonization of the respiratory tract by Pseudomonas aeruginosa are associated with a poor prognosis. Current guidelines for referral to a lung transplant center include age, sex, forced expiratory volume at one second (FEV1) below 30% predicted or a rapid decline of FEV1, in particular in young female patients, increasing frequency of exacerbations requiring antibiotic therapy, refractory or recurrent pneumothorax, recurrent hemoptysis not controlled by embolization. But, despite these criteria, near that 30% of patients are still dying while on the lung transplant waiting list, or are transplanted in high emergency. Cardiopulmonary exercise testing (CPET) in CF patients would have an interest in the following of cystic fibrosis patients. A previous study, carried out on fifty one adult patients, showed that CPET with blood gas analysis may have a prognosis value in cystic fibrosis. The authors found that a BMI < 19.8 and P(A-a)O2 peak > 43 mmHg were independently associated with a lower chance of survival.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 15 years
* Cystic fibrosis diagnosed by positive sweat chloride test or genetic test

Exclusion Criteria:

* Pregnant or breastfeeding woman
* waiting on transplantation list

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2012-03-05 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2019-06-16 (Actual)

PRIMARY OUTCOMES:
Survival | at five years
  the survival is defined by the occurrence of death or lung transplantation.

SECONDARY OUTCOMES:
6 minute walking distance | Every 12 months during 5 years
body mass index calculation | Every 12 months during 5 years
sputum sample culture | Every 12 months during 5 years
  (a descriptive analysis of Haemophilus influenzae, Staphylococcus aureus, Pseudomonas aeruginosa,Burkholderia cepacia streptococci in the bacterial flora of sputum)
pulmonary function testing with DLCO | Every 12 months during 5 years
  diffusing lung capacity for carbon monoxide.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Prevotat, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Calmette, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No